CLINICAL TRIAL: NCT07149363
Title: Adjuvant Chemotherapy and Immunotherapy for Completely Resected Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFT-61
Record Dates: First submitted 2025-08-28; First posted 2025-09-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Small Cell Lung Cancer (SCLC)
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab and one of the two chemotherapy combinations: cisplatin or carboplatin, and etoposide (Experimental): 65 participants will be enrolled.
  Interventions: Drug: Durvalumab 50 MG/ML

INTERVENTIONS:
Drug: Durvalumab 50 MG/ML — Following surgical removal of their small-cell lung cancer, participants will receive a combination of 1500 mg durvalumab and cisplatin 75 mg/m2 or carboplatin AUC 5 on day 1, and etoposide 100 mg/m2 on days 1, 2, and 3, every 3 weeks for 4 cycles (a total of 12 weeks). Following the combination of chemotherapy and immunotherapy, participants will then receive 1500 mg durvalumab every 4 weeks for 9 cycles (a total of 36 weeks).
  Other Names: Imfinzi®; MEDI4736

SUMMARY:
This is a phase II trial of adjuvant chemotherapy and immunotherapy for completely resected small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
This is a phase II open-label, single-arm, multi-center study to evaluate the efficacy and safety of adjuvant immunotherapy with chemotherapy for completely resected pathologic T1-T2, N0-N1, M0 small cell lung cancer (SCLC). The statistical design includes a predefined range of alpha and power to detect an improvement in 2-year disease free survival (DFS).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Body weight >30 kg.
* Must have a life expectancy of at least 12 weeks.
* Must have histologically or cytologically confirmed diagnosis of pathologic T1-T2 N0-1 M0 small-cell lung cancer per the American Joint Committee on Cancer staging system, 8th edition.
* Have completely resected (wedge resection, segmentectomy, lobectomy, sleeve lobectomy, bilobectomy, or pneumonectomy) small-cell lung cancer within 78 days of enrollment.
* Complete mediastinal lymph node dissection (MLND) or systematic mediastinal lymph node sampling is required.
* No prior systemic therapies, for small cell lung cancer.
* Post-operative radiation for the resected small cell lung cancer is acceptable per treating physician in the setting of N1 disease, but no other prior radiation for small cell lung cancer.
* ECOG performance status 0-1.

Exclusion Criteria:

* Patients who are receiving any other investigational agents.
* Concurrent enrollment in another clinical study involving investigational treatment directed to treatment of patients with small cell lung cancer.
* Prior treatment with durvalumab.
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of IP and of low potential risk for recurrence.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Superficial bladder cancer without active disease after treatment.
  * Low grade prostate cancer without indication for active treatment.
  * Adequately treated carcinoma in situ without evidence of disease.
* Patients with a history of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or insufficiently treated deep venous thrombosis (DVT) within the past 3 months.
* Patients with hemoptysis in excess of 2.5 mL within 2 weeks prior to the first dose of study medication.
* Patients requiring concomitant therapy with phenytoin, phenobarbital, or carbamazepine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | 2 years
  To determine whether the addition of durvalumab to adjuvant chemotherapy after surgery for limited-stage SCLC leads to improved disease free survival (DFS) when compared to historical data of participants who received adjuvant chemotherapy without immunotherapy after surgery for SCLC. DFS is measured in months from the time of surgery.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  To determine whether the addition of durvalumab to adjuvant chemotherapy after surgery for limited-stage SCLC leads to improved overall survival (OS) when compared to historical data of participants who received adjuvant chemotherapy without immunotherapy after surgery for SCLC. OS is measured in months from the time of surgery.
Safety of the regimen | 1 year
  The frequency of grade 3+ treatment-related adverse events will be reported.
Safety of the regimen | 5 years
  The frequency of grade 3+ all-cause adverse events will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Fu Jeffrey Yang, MD, Study Chair — Massachusetts General Hospital; Jacob Sands, MD, Study Chair — Dana-Farber Cancer Institute; Evanthia Galanis, MD, Principal Investigator — Alliance Foundation Trials, LLC.